CLINICAL TRIAL: NCT02511990
Title: A Phase 1, Open Label, Dose-escalation Study of the Safety, Pharmacokinetics and Antiretroviral Activity of 10-1074 Monoclonal Antibody in HIV-infected and HIV-uninfected Individuals
Brief Title: A Study of the Safety, Pharmacokinetics and Antiretroviral Activity of 10-1074
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCA-0885
Record Dates: First submitted 2015-07-24; First posted 2015-07-30 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Healthy; HIV
Keywords: HIV; 10-1074; Monoclonal Antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group 1A (Experimental): HIV-infected individuals Off ART, HIV-1 viral load < 100,000 copies/ml or On ART, HIV-1 viral load < 500 copies/ml
  3 mg/kg, single dose IV administration of 10-1074
  Interventions: Biological: 3 mg/kg, single dose IV administration of 10-1074
- Group 1B (Experimental): HIV-infected individuals Off ART, HIV-1 viral load < 100,000 copies/ml or On ART, HIV-1 viral load < 500 copies/ml
  10 mg/kg, single dose IV administration of 10-1074
  Interventions: Biological: 10 mg/kg, single dose IV administration of 10-1074
- Group 1C (Experimental): HIV-infected individuals Off ART, HIV-1 viral load < 100,000 copies/ml or On ART, HIV-1 viral load < 500 copies/ml
  30 mg/kg, single dose IV administration of 10-1074
  Interventions: Biological: 30 mg/kg, single dose IV administration of 10-1074
- Group 1D (Experimental): HIV-infected individuals Off ART, HIV-1 viral load < 100,000 copies/ml
  30 mg/kg, single dose IV administration of 10-1074
  Interventions: Biological: 30 mg/kg, single dose IV administration of 10-1074
- Group 2A (Experimental): HIV-uninfected individuals
  3 mg/kg, single dose IV administration of 10-1074
  Interventions: Biological: 3 mg/kg, single dose IV administration of 10-1074
- Group 2B (Experimental): HIV-uninfected individuals
  10 mg/kg, single dose IV administration of 10-1074
  Interventions: Biological: 10 mg/kg, single dose IV administration of 10-1074
- Group 2C (Experimental): HIV-uninfected individuals
  30 mg/kg, single dose IV administration of 10-1074
  Interventions: Biological: 30 mg/kg, single dose IV administration of 10-1074
- Group 2D (Experimental): HIV-uninfected individuals
  30 mg/kg, single dose IV administration of 10-1074
  Interventions: Biological: 30 mg/kg, single dose IV administration of 10-1074

INTERVENTIONS:
Biological: 3 mg/kg, single dose IV administration of 10-1074 — 3 mg/kg, single dose IV administration of 10-1074
  Arms: Group 1A; Group 2A
Biological: 10 mg/kg, single dose IV administration of 10-1074 — 10 mg/kg, single dose IV administration of 10-1074
  Arms: Group 1B; Group 2B
Biological: 30 mg/kg, single dose IV administration of 10-1074 — 30 mg/kg, single dose IV administration of 10-1074
  Arms: Group 1C; Group 1D; Group 2C; Group 2D

SUMMARY:
This is a phase 1 clinical trial to evaluate the safety, pharmacokinetics and the antiretroviral effects of the highly neutralizing anti-HIV-1 monoclonal antibody 10-1074 in HIV-infected and HIV-uninfected individuals.

DETAILED DESCRIPTION:
In preclinical studies carried out in humanized mice and non-human primates, 10-1074 alone or in combination with other neutralizing antibodies led to protection from HIV or simian/human immunodeficiency virus (SHIV) infection and also to sustained suppression of HIV plasma viremia. The aims of this protocol are to evaluate the safety, tolerability and pharmacokinetics profile of 10-1074 in both HIV-infected and HIV-uninfected individuals, and its antiretroviral activity in HIV-infected individuals.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (HIV-infected)

* Males and females, age 18 to 65
* HIV-1 infection confirmed by two independent assays.
* Group (1A-1C): HIV-infected individuals off ART for at least 8 weeks with HIV-1 plasma RNA levels < 100,000 copies/ml by standard assays, or on ART with HIV-1 plasma RNA levels < 500 copies/ml. HIV-1 RNA levels should be measured on 2 occasions, at least 1 week apart and one measurement must be performed within 49 days prior to enrollment.
* Group (1D): HIV-infected individuals off ART for at least 8 weeks with HIV-1 plasma RNA levels < 100,000 copies/ml by standard assays, measured on 2 occasions, at least 1 week apart. At least one measurement must be performed within 49 days prior to enrollment.
* Current CD4 count > 300 cells/μl.
* If sexually active male or female, and participating in sexual activity that could lead to pregnancy, agrees to use two effective methods of contraception from 10 days prior to the 10-1074 infusion until the end of the study.

Group 2 (HIV-uninfected):

* Males and females, age 18 to 65.
* Amenable to HIV risk reduction counseling and agrees to maintain behavior consistent with low risk of HIV exposure.
* If sexually active male or female, and participating in sexual activity that could lead to pregnancy, agrees to use two effective methods of contraception throughout the study period, as described for the HIV-infected groups above.

Exclusion Criteria:

Group 1 (HIV-infected):

* Have a history of AIDS-defining illness within 1 year prior to enrollment.
* History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months.
* Any clinically significant acute or chronic medical condition other than HIV infection, that in the opinion of the investigator would preclude participation.
* Chronic Hepatitis B or Hepatitis C infection.
* Laboratory abnormalities in the parameters listed below:

Absolute neutrophil count ≤ 1,000; Hemoglobin ≤10 gm/dL; Platelet count ≤100,000; ALT ≥ 2.0 x ULN; AST ≥ 2.0 x ULN; Total bilirubin ≥ 1.25 x ULN; Creatinine ≥ 1.1 x ULN; Coagulation parameters (PT, PTT or INR) ≥ 1.25 x ULN.

* Pregnancy or lactation.
* Any vaccination within 14 days prior to 10-1074 administration.
* History of severe reaction to a vaccine or drug infusion or history of severe allergic reactions.
* Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.

Group 2 (HIV-uninfected):

* Confirmed HIV-1 or HIV-2 infection.
* History of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months.
* Any clinically significant acute or chronic medical condition (such as autoimmune diseases) that in the opinion of the investigator would preclude participation.
* Within the 12 months prior to enrollment, the volunteer has a history of sexually transmitted infection.
* Chronic Hepatitis B or Hepatitis C infection.
* Laboratory abnormalities in the parameters listed:

Absolute neutrophil count ≤ 1,500; Hemoglobin ≤ 12 gm/dL if female; ≤ 13.5 gm/dL if male; Platelet count ≤ 140,000; Alanine transaminase (ALT) ≥ 1.25 x upper limit of normal (ULN); aspartate transaminase (AST) ≥ 1.25 x ULN; Total bilirubin ≥ 1.25 x ULN; Creatinine ≥ 1.1 x ULN; Coagulation parameters (prothrombin time - PT, partial thromboplastin time - PTT or INR) ≥ 1.25 x ULN.

* Pregnancy or lactation.
* Any vaccination within 14 days prior to 10-1074 administration.
* Receipt of any experimental HIV vaccine in the past.
* History of severe reaction to a vaccine or drug infusion or history of severe allergic reactions.
* Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 weeks after 10-1074 administration

SECONDARY OUTCOMES:
Serum peak concentration of 10-1074, measured in micrograms per ml | 24 hours after 10-1074 administration
Serum half-life of 10-1074 expressed in days | 24 Weeks after 10-1074 administration
Plasma HIV-1 RNA levels measured in copies/ml | 2 weeks after 10-1074 administration

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — Rockefeller University
Locations (2):
- The Rockefeller University, New York, New York, United States
- University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No